CLINICAL TRIAL: NCT05495594
Title: Central Sensitization and Releated Factors in Medical Students: a Cross-Sectional Study
Brief Title: Central Sensitization in Medical Students
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Nihan ERDINC GUNDUZ, assistant professor,MD, Dokuz Eylul University
Other Study IDs: TıpFakogrencisantralsensitzsyn
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Central Sensitisation
Keywords: Central Sensitisation; medical students; Central Sensitisation inventory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Central sensitization (SS); is a physiological phenomenon caused by neuronal dysregulation and hyperexcitability in the central nervous system, resulting in hypersensitivity to painful and painless stimuli.Central sensitization syndromes (CSS); defines disorders in which SS originates and cannot be medically explained by any organic cause. CSS include clinical conditions such as fibromyalgia syndrome (FMS), chronic fatigue syndrome (CFS), temporomandibular joint disorders (TMD), migraine/tension type headache, irritable bowel syndrome (IBS), restless legs syndrome (RLS). These disorders have many common clinical features such as pain, fatigue, sleep disturbance, increased sensitivity to painful and painless stimuli, coexistence, paresthesia, psychosocial disorders, and show the presence of SS.

The Central Sensitization Inventory (SSI) is a short, easy-to-apply scale consisting of 25 questions that identifies key symptoms in patients with SS and quantifies the degree of these symptoms. The Turkish adaptation and validity-reliability study of the SSE was conducted in 2021.

In this descriptive, cross-sectional study, it was planned to investigate the presence of central sensitization and related factors in medical faculty students.

In the 2021-2022 academic year of Dokuz Eylul University Faculty of Medicine, a total of 324 students, the number determined as a result of power analysis, will be asked to fill in a short form in which the factors related to the "Central Sensitization Inventory" and demographic data are questioned. Then, statistical analysis will be applied with the analyzed data.In addition, Central Sensitization Inventory scores of students in each term will be compared with each other.

DETAILED DESCRIPTION:
Central sensitization (SS); It is a physiological phenomenon caused by neuronal dysregulation and hyperexcitability in the central nervous system, resulting in hypersensitivity to painful and painless stimuli. It is characterized by abnormal pain increase due to neuronal hyperreactivity and dysfunction of the descending and ascending pathways. The hypersensitivity state of the central nervous system develops due to the amplification of neuronal signals with various synaptic and neurotransmitter activities, regardless of defined peripheral inputs.

It was first described by Woolf in 1983 based on studies showing that spinal neuron hyperexcitability can be induced by peripheral tissue damage in rats. Central sensitization syndromes (CSS); it defines disorders in which SS originates and cannot be medically explained by any organic cause. CNS include clinical conditions such as fibromyalgia syndrome (FMS), chronic fatigue syndrome (CFS), temporomandibular joint disorders (TMD), migraine/tension type headache, irritable bowel syndrome (IBS), restless legs syndrome (RLS). These disorders have many common clinical features such as pain, fatigue, sleep disturbance, increased sensitivity to painful and painless stimuli, co-occurrence, paresthesia, psychosocial disorders, and show the presence of SS.

Other factors that may or may not be associated with SS; genetics, excessive sympathetic activity, endocrine dysfunction (e.g. hypofunction of the adrenal cortex and decreased growth hormone), poor sleep quality, viral infection, peripheral nociceptive sources (e.g. arthritis), environmental stimuli (air, light, noise, etc.), childhood bad experiences and psychosocial disorders.

The Central Sensitization Inventory (SSI) is a short, easy-to-apply scale consisting of 25 questions that identifies key symptoms in those with SS and quantifies the degree of these symptoms. It was developed in 2012. It helps to distinguish between different types of chronic pain patients with different degrees of SS, and makes it easier to distinguish whether the pain is due to organic causes or central sensitization.

The SSI consists of 2 parts, part A, which evaluates the symptoms thought to be associated with SS syndromes, and part B, which quickly questions whether the patient has previously received a specific diagnosis. Part A of the SSE includes all CNS symptoms, which will help clinicians identify the CNS patient. In part A, there are 25 items that question the frequency of symptoms seen in SS syndromes and are scored between 0-100 points. Each symptom is defined as "never" (0 points) if the patient never experiences that symptom, "rarely" (1 point) if rarely, "sometimes" if sometimes (2 points), "frequently" if experienced frequently (3 points), if experienced always, it is recorded as "always" (4 points). It is accepted that SS develops in those who score above 40 on the scale. As the patient's SSI score increases, it is thought that he has more SS-related symptoms. In addition, the B part of the scale (no scoring) is the part that includes 7 separate parts that asks whether he has received any diagnosis related to one or more CNS or related conditions.

With this scale, it is aimed to help clinicians better evaluate the symptoms thought to be associated with SS, to minimize or, if possible, prevent unnecessary diagnostic and treatment procedures. The Turkish adaptation and validity-reliability study of the SSI was conducted in 2021.

In this descriptive, cross-sectional study, it was planned to investigate the presence of central sensitization and related factors in Medical Faculty students. In the 2021-2022 academic year of Dokuz Eylul University Faculty of Medicine, a total of 324 students, the number determined as a result of power analysis, will be asked to fill in a short form in which the factors related to the "Central Sensitization Inventory" and demographic data are questioned.

Power analysis was done with Openepi program. In the Openepi program, it is planned to reach at least 324 students at a 95% confidence level, with a margin of error of 50% and 5% as the worst, for 80% power over 2038 total number of students.

Distribution was made according to classes by calculation with stratified sampling method. It is planned to include at least 59 students for Term 1, at least 51 for Term 2, at least 55 for Term 3, at least 54 for Term 4, at least 47 for Term 5, and at least 59 for Term 6

Then, statistical analysis will be applied with the analyzed data. In addition, Central Sensitization Inventory scores and releated factors of students in each term will be compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being a medical student

Exclusion Criteria:

* neurological disease
* rheumatic disease
* uncontrolled hypothyroidism
* hyperparathyroidism
* diabetes mellitus
* infectious diseas
* malignancy
* not signing the voluntary consent form

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Medical students aged between 18-25 years old
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The Central Sensitization Inventory | baseline
  The Central Sensitization Inventory consists of 2 parts, part A and B.In part A, there are 25 items that question the frequency of symptoms seen in SS syndromes and are scored between 0-100 points. Each symptom is defined as "never" (0 points) if the patient never experiences that symptom, "rarely" (1 point) if rarely, "sometimes" if sometimes (2 points), "frequently" if experienced frequently (3 points), if experienced always, it is recorded as "always" (4 points). It is accepted that SS develops in those who score above 40 on the scale (3). As the patient's SSI score increases, it is thought that he has more SS-related symptoms. In addition, the B part of the scale (no scoring) is the part that includes 7 separate parts that asks whether he has received any diagnosis related to one or more CNS or related conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Akalın, MD,Prof, Study Director — Medical Faculty of Dokuz Eylül University, İzmir, Turkey
Locations (1):
- 1Department of Physical Medicine and Rehabilitation, Medical Faculty of Dokuz Eylül University, İzmir, Turkey, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Background] Yunus M. Central sensitivity syndromes: a unified concept for fibromyalgia and other similar maladies. J Indian Rheum Assoc 2000;8(1):27-33
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Duzce Keles E, Birtane M, Ekuklu G, Kilincer C, Caliyurt O, Tastekin N, Is EE, Ketenci A, Neblett R. Validity and reliability of the Turkish version of the central sensitization inventory. Arch Rheumatol. 2021 Oct 18;36(4):518-526. doi: 10.46497/ArchRheumatol.2022.8665. eCollection 2021 Dec. PMID 35382371
- [Background] Kindler LL, Bennett RM, Jones KD. Central sensitivity syndromes: mounting pathophysiologic evidence to link fibromyalgia with other common chronic pain disorders. Pain Manag Nurs. 2011 Mar;12(1):15-24. doi: 10.1016/j.pmn.2009.10.003. Epub 2009 Dec 2. PMID 21349445
- [Background] Yunus MB. Fibromyalgia and overlapping disorders: the unifying concept of central sensitivity syndromes. Semin Arthritis Rheum. 2007 Jun;36(6):339-56. doi: 10.1016/j.semarthrit.2006.12.009. Epub 2007 Mar 13. PMID 17350675
- [Background] Woolf CJ, Thompson SW, King AE. Prolonged primary afferent induced alterations in dorsal horn neurones, an intracellular analysis in vivo and in vitro. J Physiol (Paris). 1988-1989;83(3):255-66. PMID 3272296
- [Background] Aaron LA, Buchwald D. A review of the evidence for overlap among unexplained clinical conditions. Ann Intern Med. 2001 May 1;134(9 Pt 2):868-81. doi: 10.7326/0003-4819-134-9_part_2-200105011-00011. PMID 11346323
- [Background] McBeth J, Macfarlane GJ, Benjamin S, Morris S, Silman AJ. The association between tender points, psychological distress, and adverse childhood experiences: a community-based study. Arthritis Rheum. 1999 Jul;42(7):1397-404. doi: 10.1002/1529-0131(199907)42:73.0.CO;2-7. PMID 10403267